CLINICAL TRIAL: NCT06171425
Title: Diffüz Parankimal Akciğer Hastalarında Kırılganlık Düzeyi, Egzersiz Kapasitesi ve Denge Değerlendirilmesi
Brief Title: Evaluation of Patients With Diffuse Parenchymal Lung Diseases Regarding Frailty
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Aynur Demirel, PT, PhD, Assoc. Prof., Hacettepe University
Other Study IDs: GO 23/18
Record Dates: First submitted 2023-10-30; First posted 2023-12-14 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Diffuse Parenchymal Lung Disease; Frailty; Physical Inactivity
MeSH Terms: conditions — Lung Diseases, Interstitial; Frailty; Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DPAH group: patients with diffuse parenchymal lung diseases
- control group: aged matched healthy patients

SUMMARY:
There are very few studies in the literature examining the frailty levels of diffuse parenchymal lung disease (DPLD) patients and its effect on their functional status despite the high prevalance of frailty in patients with DPLD This observational study aims to learn about the relationship between frailty and functional capacity and balance in DPLD patients compared to healthy subjects.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the relationship between the level of frailty and exercise capacity, respiratory functions, diffusion capacity, balance level, postural changes, activities of daily living, peripheral muscle strength and quality of life parameters in DPLD patients. The second aim is to compare diffuse parenchymal lung patients and the healthy control group in terms of these parameters.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with Diffuse parenchymal lung according to the American Thoracic Society/European Respiratory Society (ATS/ERS) criteria,
* Being between the ages of 30-65,
* Being literate,
* Being willing to participate in the research,
* Being clinically stable and having any accompanying comorbid conditions (such as hypertension, diabetes) under control,
* Not having any orthopedic, metabolic or neurological problems that may prevent evaluation of peripheral muscle strength, balance and exercise capacity.

Exclusion Criteria:

* Having recently experienced syncope,
* Having a history of unstable cardiovascular disease,
* Having been hospitalized due to exacerbation in the last 3 months,
* Having received pulmonary rehabilitation in the last 12 months,
* Having a neurological disease,
* Being dependent and using a walking aid while performing the person's daily life activities,
* Having a pacemaker,
* Having a diagnosis of lung cancer

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred by the department of chest diseases of Hacettepe university will be taken
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-12-25 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-22 (Estimated)

PRIMARY OUTCOMES:
frailty level | 1 time which will be in one day
  evaluation of frailty level with Fried Frailty Criteria which are weight loss existence, muscle strength, physical activity (will be measured with International Physical Activity Questionnaire), mobility (will be measured by 4-meter walking test), and depression level. Fried frailty phenotype consists of five criteria: loss, exhaustion, physical inactivity, low hand grip strength, and slow walking speed. Patients who have three or more of these criteria are defined as frail, those who have one or two criteria, are defined as prefrail, and none of the criteria are defined as robust.

SECONDARY OUTCOMES:
comorbidity assesment | 1 time which will be in one day
  via Charlson comorbidity index (values between 0-33)
exercise capacity | 1 time which will be in one day
  by 1 minute sit to stand test
balance measurement | day 1
  by timed up and go test
posture analysis | day 1
  corbin postural assesment scale from lateral and posterior view will be applied. The Corbin Posture Scale is a postural assessment scale that evaluates the inclination of the head in different directions, the shape of the dorsal region, the presence of scapulaand shoulder protraction, the signs of scoliosis, kyphosis, lordosis, whether there is a difference in the height of the two shoulders and hips, the sagging status in the abdominal region, the presence of gibbosity, genu recurvatum, and the level of anterior balance by assigning a score between 0-3.
posture related conditions measurement | day 1
  observational analysis by scapular dyskinesia test
posture related (scapular motion)conditions existence measurement | day 1
  by lateral scapular slide test which evaluates distance between medial border of spine scapulae and T3 spinous process- T7 spinous process and inferior angle of scapulae
quality of life evaluation | day 1
  Quality of life will be assessed by Saint George respiratory questionnaire. A total score is calculated from 0 (no health impairment) to 100 (maximum health impairment).
evaluation of participation to daily life activities | day 1
  Participation to daily life activities will be evaluated by London Chest Activities of Daily Living Questionnare. Contains 15 items grouped into four domains: self-care, household activities (domestic), physical, and leisure activities. Responses for each item range from 0-5, with 0 indicating "wouldn't do anyway", 1-4 representing degree of breathlessness and 5 representing the greatest difficulty with performing ADL (someone else completes). Responses to items 1-15 are added; the total score can range from 0 to 75 points, with higher scores indicating greater functional limitation
pulmonary function measurement | day 1
  evaluation of pulmonary function with lung function test which will be detected via FVC, FEV1, FEV1/FVC, PEF, FEF25-75% At least three technically acceptable measurements were obtained between the two best-measured FEV1 values, with no more than a 5% difference, and the best FEV1 value was selected for analysis.
investigation of diffusion capacity of the lung | day 1
  by diffusion capacity of carbon monoxide of lung with single breath method
peripheral muscle strength | day 1
  by hand held dynamometry device

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Health Sciences Faculty, Ankara, Turkey (Türkiye)